CLINICAL TRIAL: NCT04367389
Title: Internet-based Physical Activity Promotion and Exercise Prescription for People With Multiple Sclerosis
Acronym: ms bewegt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Neurological Rehabilitation Center Quellenhof (Unknown); ZTM Bad Kissingen (Other); Medi train - Zentrum für Gesundheitssport, Sport- und Physiotherapie (Unknown); proMX GmbH Nürnberg (Unknown); motionNET systems Limited (Unknown); Aktion Multiple Sklerose Erkrankter, Landesverband der DMSG in Baden-Württemberg (AMSEL) e.V. (Unknown); Klinikum Würzburg Mitte GmbH (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Head of the Department of Sport Science and Sport, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ms bewegt 2.0
Record Dates: First submitted 2020-04-21; First posted 2020-04-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; physical activity; exercise; behavior change; internet-based intervention; physical literacy; self-determination theory
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive a physical activity promotion intervention as well as an individualized exercise plan.
  Interventions: Behavioral: Physical activity promotion; Behavioral: Exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity promotion — Physical activity promotion activities consist of two phone or video calls with a therapists, two group video calls with a therapist, a complementary e-learning course and a fitness tracker that was provided.
  Arms: Intervention
Behavioral: Exercise — Participants will agree with their therapist on an exercise plan (endurance and resistance training) that will be made available through the studies mobile app. Frequency and duration of endurance and strength training shall be prescribed in accordance with exercise guidelines for persons with MS. However, they can be adjusted according to participants prior physical activity level and their time for exercise during the week.
  Arms: Intervention

SUMMARY:
The aim of the study is to evaluate the effects of a 12-week internet-based exercise and physical activity promotion intervention on physical activity. Furthermore, effects on symptoms of Multiple Sclerosis, Physical Activity-related Health Competence (PAHCO), self-concordance and basic needs satisfaction as well as usability and acceptability of the intervention will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed Multiple Sclerosis (McDonald criteria)
* Expanded Disability Status Scale between 0 - 6.5
* neurologically stable (no exacerbation within 30 days prior to enrollment)
* internet access (WiFi)
* basic knowledge on handling personal computer and the internet
* owning a smartphone with the operating system Android or IOS and with access to Google Play Store or Apple App score
* basic computer and internet skills (e. g. using web browser and webcams)
* ability to operate a smartphone (especially to install mobile applications)
* ability to read, write and comprehend as well as communicate electronically

Exclusion Criteria:

* regularly physically active (more than 30 minutes twice a week with at least moderate intensity; includes aerobic training, resistance training and other sports e.g. Tennis; excludes physiotherapy, physical activity during work or household, grocery shopping, gardening, walking the dog etc.)
* clinically relevant cardiovascular diseases
* cortisone therapy in the last 30 days
* cognitive impairment that hampers study implementation
* severe impairment of hand function (ataxia or paresis impeding the use of a smartphone app or smartwatch)
* severe internal, orthopaedic and metabolic diseases that restrict mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in objectively measures physical activity | Baseline, after 3 months, after 6 months
  The physical activity level of participants is measured over a 7 day period with the accelerometer Actigraph GT3X+. The Actigraph GT3X+ measures acceleration on three axes. Steps per day, physical activity per day (activity counts) and time in moderate and vigorous physical activity per day will be calculated.

SECONDARY OUTCOMES:
Changes in subjectively measured physical activity: BSA-Questionnaire | Baseline, after 3 months, after 6 months
  The questionnaire asks for physical activities during a typical week. It differentiates between leisure-time/transportation activities (physical activity score) and sport-/exercise-related activities (sports score). Participants are required to report frequency and duration of activities executed during the last two weeks. Minutes of leisure-time physical activity per week and sport-/exercise related activity per week are calculated to get the physical activity and the sports score. Both scores can combined in order to receive the overall volume of physical activity completed during leisure-time and transportation as well as sport-/exercise-related activities.
Würzburger Fatigue Inventory for MS (WEIMuS) | Baseline, after 3 months, after 6 months
  This questionnaire contains 17 items that form a physical and cognitive subscale. The total score ranges from zero to a maximum of 68 points (maximum fatigue). The cut-off value for the presence of fatigue is above 32.
Allgemeine Depressionsskala (ADS-L) | Baseline, after 3 months, after 6 months
  German version of the Center for Epidemiologic Studies Depression Scale, 20 item questionnaire. Each item is rated on a 4-point Likert scale. Answers are scored from 0 to 3. The scores for all items are added up to receive the total score. The total score ranges from 0 to 60 with higher scores representing higher levels of depression.
Multiple Sclerosis Walking Scale-12 | Baseline, after 3 months, after 6 months
  12-item questionnaire measuring self reported walking ability. Each item is answered on a 5-point Likert scale. Answers are scored from 1 to 5. The scores for all items are added up to receive a total score. The total score ranges from 12 to 60 with higher scores representing higher levels of depression. As a last step the total score is transformed into the walk12-score ranging from 0 to 100 ((total score -12)/48 x 100 = walk12-score).
Multiple Sclerosis Impact Scale (MSIS-29) | Baseline, after 3 months, after 6 months
  An disease-specific questionnaire that measures quality of life and limitations due tu multiple sclerosis on two subscales (physical impact of MS, 20 items; psychological impact of MS, 9 items).Scores for both scales are generated by summing individual item scores and transforming the sum to a 0-100 scale. Higher scores represent worse health.
Timed 25-Foot Walk Test (T25FW) | Baseline, after 3 months, after 6 months
  The task is to walk a 25foot distance as fast as possible. This test measures the functionality of the lower extremity and the walking speed.
Two-minute Walk Test (2MWT) | Baseline, after 3 months, after 6 months
  The 2MWT measures walking endurance. It measures walking distance over 2 minutes. The subject is asked to walk as far as possible in 2 minutes.
Selbstkonkordanz-Skala (SSK-Scale) | Baseline, after 3 months, after 6 months
  The SSK-Scale measures self-rated physical activity-related and sports-related self-concordance. It contains 12 items which are assigned to 4 subscales: intrinsic, identified, introjected and extrinsic Motivation. An overall score can be calculated based on these four subscales (minimal score = -10, maximal Score = +10). To receive the overall score the scores of the subscales for introjected and extrinsic motivation will be subtracted from the sum of the identified and intrinsic motivation subscales. A high total score suggest a high level of physical activity-related and sports-related self-concordance.
Physical activity-related health competence questionnaire | Baseline, after 3 months, after 6 months
  44-item questionnaire that measures physical activity-related health competence. The physical activity related health competence consists of three subcompetencies: movement competence (20 items; min = 0, max = 17.6), control competence (10 items; min = 0, max = 10.8), PA-related self-regulation competence (14 items; min = 0, max = 14.8).
German psychological need satisfaction in exercise scale | Baseline, after 3 months, after 6 months
  This is a questionnaire to estimate the satisfaction of the three basic psychological needs based on self-determination theory during sports- and exercise related activities. It consists of 11 items which are assigned to 3 scales (one for each psychological need). Higher values on the scales indicate a higher needs satisfaction.
Usability and usefulness of the mobile application (meCue 2.0 questionnaire) | after 3 months, after 6 months
  The module usability and usefulness of the meCue 2.0 questionnaire was used. The module contains 3 items on usability and 3 items on usefulness that are answered on a 7-point Likert scale (scored from 1 to 7). In order two receive a score for usability and a score for usefulness, the mean is calculated for the items of each area.
Usability and usefulness of the intervention | after 3 months, after 6 months
  Questionnaire including the Net Promoter Score and 45 self-developed items. Self-developed items covered willingness to pay, goal attainment, effects on physical function and wellbeing, adequacy of exercise prescription, evaluation of communication within the program, learning modules, App functions and activity trackers.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander University Erlangen-Nürnberg; Peter Flachenecker, Prof. Dr. med., Principal Investigator — Neurological Rehabilitation Center Quellenhof; Mathias Mäurer, Prof. Dr. med., Principal Investigator — Klinikum Würzburg Mitte gGmbH
Locations (9):
- Germany (9):
  - Neurological Rehabilitation Center Quellenhof, Bad Wildbad
  - Friedrich-Alexander University Erlangen-Nürnberg, Erlangen
  - Kliniken Schmieder Konstanz, Konstanz
  - Facharztpraxis für Neurologie und Psychiatrie Dr. med Wolfgang Mattes und Andreas Stockert, Pforzheim
  - Fachklinik für Neurologie Dietenbronn GmbH, Schwendi
  - E/M/S/A - Zentrum für Neurologie/Psychiatrie/Neuroradiologie, Singen
  - Klinikum Stuttgart Katharinenhospital, Stuttgart
  - Neurologisch-Psychiatrische Praxis Dr. Weber, Stuttgart
  - Klinikum Würzburg Mitte gGmbH, Würzburg

REFERENCES:
- [Derived] Hartung V, Tallner A, Flachenecker P, Maurer M, Streber R, Wanner P, Rashid A, Shammas L, Hois G, Dettmers C, Roick H, Stefanou A, Tumani H, Weber S, Pfeifer K. Internet-based exercise and physical activity promotion for persons with multiple sclerosis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Apr 23;17(1):90. doi: 10.1186/s13102-025-01146-x. PMID 40270018